CLINICAL TRIAL: NCT04581421
Title: The Role of Dietary Carbohydrate and Fat Availability in the Regulation of Hepatic Lipid Content
Acronym: LICARB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Danish Research Centre for Magnetic Resonance (Other)
Responsible Party: Principal Investigator, Kirstine Nyvold Bojsen-Moeller, Principal investigator, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LICARB ID PhD010-19.
Record Dates: First submitted 2020-09-25; First posted 2020-10-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: NAFLD; Overweight and Obesity; Metabolic Syndrome; Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight; Obesity; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized diet intervention study in a cross over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Carb first (Experimental)
  Interventions: Other: High Carb Low Fat Diet; Other: Low Carb High Fat Diet
- Low Carb first (Experimental)
  Interventions: Other: High Carb Low Fat Diet; Other: Low Carb High Fat Diet

INTERVENTIONS:
Other: High Carb Low Fat Diet — The participants will be randomized to a diet of low carb/ high fat og high carb/low fat
Other: Low Carb High Fat Diet — The participants will be randomized to a diet of low carb/ high fat og high carb/low fat

SUMMARY:
The purpose of this study is to investigate dietary compositions effect on liverfat measured by magnetic resonance imaging.

DETAILED DESCRIPTION:
Overweight but otherwise healthy men will be included in the study which is a randomized diet intervention study in a cross over design.

The study involves 2 intervention periods of 5 days each, during which the participant ingests two different types of experimental diet. Participants will in randomized order (determined by block randomization) ingest a diet with low carbohydrate and high fat content, and a diet with high carbohydrate and low fat content.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men being 18-50 years old.
* Overweight (BMI 25-35)
* Low to moderate physical activity level, defined as ≤ 1 weekly session of aerobic exercise.
* Non-smokers
* No use of medicine

Exclusion Criteria:

* Fasting blood glucose indicating overt diabetes (≥7 mmol/l)
* HbA1C >48 mmol/mol
* Fasting plasma triacylglycerol indicating dyslipidemia (≥2.2 mmol/l)
* FIB-4 score >1.45
* Contraindications for MR-scan: abdominal height exceed limitations of the MR-scanner, pacemaker or other electronic device implanted, implanted metal devices, severe claustrophobia.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Liverfat | (MRS Day -1 (before intervention starts), Day 5 (after diet intervention is completed)
  The effect of high-carbohydrate/low-fat vs low-carbohydrate/high-fat diet on change in MRS determined liver fat.

SECONDARY OUTCOMES:
Glycogen | (MRS Day -1 (before intervention starts), Day 5 (after diet intervention is completed)
  effect of the low-carbohydrate/high-fat intake and high-carbohydrate/low-fat intake on hepatic glycogen content measured by 7T 13C-MRS
fasting hepatic glucose output | (Day 0 and Day 6 of the diet intervention)
  measured by Ra of glucose= (infusion rate of 6,6 2H2-glucose)/TTR
fasting blood triacylglycerol concentration | (Day 0 and Day 6 of the diet intervention)
Insulin clearance determined during steady state insulin infusion | (Day 0 and Day 6 of the diet intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Amalie London, Hvidovre, Denmark

REFERENCES:
- [Derived] London A, Richter MM, Sjoberg KA, Wewer Albrechtsen NJ, Povazan M, Drici L, Schaufuss A, Madsen L, Oyen J, Madsbad S, Holst JJ, van Hall G, Siebner HR, Richter EA, Kiens B, Lundsgaard A, Bojsen-Moller KN. The impact of short-term eucaloric low- and high-carbohydrate diets on liver triacylglycerol content in males with overweight and obesity: a randomized crossover study. Am J Clin Nutr. 2024 Aug;120(2):283-293. doi: 10.1016/j.ajcnut.2024.06.006. Epub 2024 Jun 22. PMID 38914224